CLINICAL TRIAL: NCT03492281
Title: An International Phase 3, Randomized, Double-Blind, Placebo- and Active (Tolterodine)-Controlled Multicenter Study to Evaluate the Safety and Efficacy of Vibegron in Patients With Symptoms of Overactive Bladder
Brief Title: A Study to Examine the Safety and Efficacy of a New Drug in Patients With Symptoms of Overactive Bladder (OAB)
Acronym: Empowur
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Urovant Sciences GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-901-3003; 2017-003293-14 (EudraCT Number)
Record Dates: First submitted 2018-03-21; First posted 2018-04-10 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Overactive Bladder
Keywords: Beta-3 adrenergic receptor (β3-AR) agonists; Incontinence; OAB; Vibegron; Urge urinary incontinence; Urinary bladder, overactive; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Agents
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge; Urologic Diseases; Lower Urinary Tract Symptoms | interventions — N-(4-((5-(hydroxy(phenyl)methyl)pyrrolidin-2-yl)methyl)phenyl)-4-oxo-4,6,7,8-tetrahydropyrrolo(1,2-a)pyrimidine-6-carboxamide; Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vibegron + Placebo to match Tolterodine (Experimental)
  Interventions: Drug: vibegron; Drug: Tolterodine placebo
- Placebo to match vibegron + Placebo to match Tolterodine (Placebo Comparator)
  Interventions: Drug: Vibegron placebo; Drug: Tolterodine placebo
- Tolterodine + Placebo to match vibegron (Active Comparator)
  Interventions: Drug: Vibegron placebo; Drug: Tolterodine Tartrate ER

INTERVENTIONS:
Drug: vibegron — single daily oral dose of vibegron 75 mg for 12 weeks
  Other Names: RVT-901; MK4618; KRP114V; URO-901
  Arms: Vibegron + Placebo to match Tolterodine
Drug: Vibegron placebo — placebo to match vibegron (experimental drug)
  Arms: Placebo to match vibegron + Placebo to match Tolterodine; Tolterodine + Placebo to match vibegron
Drug: Tolterodine Tartrate ER — single daily oral dose of tolterodine tartrate ER 4 mg for 12 weeks
  Other Names: Mariosea XL
  Arms: Tolterodine + Placebo to match vibegron
Drug: Tolterodine placebo — placebo to match tolterodine (active comparator)
  Arms: Placebo to match vibegron + Placebo to match Tolterodine; Vibegron + Placebo to match Tolterodine

SUMMARY:
This study is designed to evaluate the safety, tolerability, and efficacy of vibegron administered once daily in patients with OAB.

ELIGIBILITY:
Inclusion Criteria:

1. Has a history of OAB for at least 3 months prior to the Screening Visit.
2. Meets either the OAB Wet or OAB Dry criteria.

Exclusion Criteria:

Urology Medical History

1. Patient had an average total daily urine volume > 3000 mL in the past 6 months or during the 14-day Run-in Period.
2. Has lower urinary tract pathology that could, in the opinion of the Investigator, be responsible for urgency, frequency, or incontinence.
3. Has a history of surgery to correct stress urinary incontinence, pelvic organ prolapse, or procedural treatments for BPH within 6 months of Screening.
4. Has current history or evidence of Stage 2 or greater pelvic organ prolapse (prolapse extends beyond the hymenal ring).
5. Patient is currently using a pessary for the treatment of pelvic organ prolapse.
6. Has a known history of elevated post-void residual volume defined as greater than 150 mL.
7. Has undergone bladder training or electrostimulation within 28 days prior to Screening or plans to initiate either during the study.
8. Has an active or recurrent (> 3 episodes per year) urinary tract infection by clinical symptoms or pre-defined laboratory criteria.
9. Has a requirement for an indwelling catheter or intermittent catheterization.
10. Has received an intradetrusor injection of botulinum toxin within 9 months prior to Screening.
11. Has uncontrolled hyperglycemia (defined as fasting blood glucose > 150 mg/dL or 8.33 mmol/L and/or non-fasting blood glucose > 200 mg/dL or 11.1 mmol/L) or, if in the opinion of the Investigator, is uncontrolled.
12. Has evidence of diabetes insipidus.
13. Is pregnant, breast-feeding, or is planning to conceive within the projected duration of the study.
14. Has a concurrent malignancy or history of any malignancy within 5 years prior to signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
15. Has uncontrolled hypertension (systolic blood pressure of ≥ 180 mmHg and/or diastolic blood pressure of ≥ 100 mmHg) or has a resting heart rate (by pulse) > 100 beats per minute.
16. Has narrow angle glaucoma (primary open angle glaucoma is not excluded).
17. Has a history of cerebral vascular accident, transient ischemic attack, unstable angina, myocardial infarction, coronary artery interventions (e.g., coronary artery bypass grafting or percutaneous coronary interventions [e.g., angioplasty, stent insertion]), or neurovascular interventions (e.g., carotid artery stenting) within 6 months prior to the Screening Visit. Has a known history of liver disease.
18. Has a history of injury, surgery, or neurodegenerative diseases (e.g., multiple sclerosis, Parkinson's) that could affect the lower urinary tract or its nerve supply.
19. Has hematuria, including microscopic hematuria according to pre-defined criteria.
20. Has clinically significant electrocardiogram (ECG) abnormality.
21. Has alanine aminotransferase or aspartate aminotransferase > 2.0 times the upper limit of normal (ULN), or bilirubin (total bilirubin) > 1.5 x ULN (or > 2.0 x ULN if secondary to Gilbert syndrome or pattern consistent with Gilbert syndrome).
22. Has an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m2.
23. Has an allergy, intolerance, or a history of a significant clinical or laboratory adverse experience associated with any of the active or inactive components of the vibegron formulation or tolterodine formulation.
24. Is currently participating or has participated in a study with an investigational compound or device within 28 days prior to signing informed consent, or has participated in any previous study with vibegron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1530 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (213):
- United States (189):
  - Central Alabama Research, Birmingham, Alabama
  - Achieve Clinical Research, Birmingham, Alabama
  - Fundamental Research LLC, Gulf Shores, Alabama
  - Longwood Research, Huntsville, Alabama
  - Coastal Clinical Research Inc., Mobile, Alabama
  - Clinical Research Consortium, Tempe, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Dream Team Clinical Research LLC, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - Core Healthcare Group, Cerritos, California
  - Research Center of Fresno Inc., Fresno, California
  - American Clinical Trials, Hawaiian Gardens, California
  - Marvel Clinical Research, Huntington Beach, California
  - Grossmont Center for Clinical Research, La Mesa, California
  - Prime-Care Clinical Research, Laguna Hills, California
  - Long Beach Clinical Trial Services Inc., Long Beach, California
  - Long Beach Clinical Trials LLC, Long Beach, California
  - Downtown L.A. Research Center Inc., Los Angeles, California
  - Urology Group of Southern California, Los Angeles, California
  - Tri Valley Urology Medical Group, Murrieta, California
  - Northern California Research, Sacramento, California
  - San Bernadino Urological Associates, San Bernardino, California
  - Artemis Institute for Clinical Research, San Diego, California
  - WR MCCCR, San Diego, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Empire Clinical Research, Upland, California
  - Bayview Research Group LLC, Valley Village, California
  - Horizons Clinical Research Center, Denver, Colorado
  - Lynn Institute of Denver, Denver, Colorado
  - Clinical Research Consulting LLC, Milford, Connecticut
  - Coastal Connecticut Research LLC, New London, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Innovative Medical Research of South Florida Inc., Aventura, Florida
  - PAB Clinical Research, Brandon, Florida
  - Innovative Research of West FL Inc., Clearwater, Florida
  - Universal Medical and Research Center LLC, Coral Gables, Florida
  - Top Medical Research Inc., Cutler Bay, Florida
  - Avail Clinical Research, DeLand, Florida
  - Jesscan Medical Research, Delray Beach, Florida
  - Revival Research, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - KO Clinical Research, Fort Lauderdale, Florida
  - A.G.A Clinical Trials, Hialeah, Florida
  - Indago Research Health Center, Hialeah, Florida
  - Best Quality Research, Inc., Hialeah, Florida
  - Vital Pharm Research Inc., Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - LCC Medical Research Institute Inc., Miami, Florida
  - Nuren Medical Research Center, Miami, Florida
  - AppleMed Research Group LLC, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Suncoast Clinical Research Inc., New Port Richey, Florida
  - Bayside Clinical Research, New Port Richey, Florida
  - Compass Research LLC, Orlando, Florida
  - South Broward Research LLC, Pembroke Pines, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - Meridien Research, Spring Hill, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Bioclinica Research, The Villages, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - In-Quest Medical Research, LLC, Peachtree Corners, Georgia
  - Meridian Clinical Research LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Evanston Premier Healthcare Research, Evanston, Illinois
  - Clinical Investigation Specialists Inc., Gurnee, Illinois
  - Investigators Research Group LLC, Brownsburg, Indiana
  - MediSphere Medical Research Center, Evansville, Indiana
  - Heartland Research Associates LLC, Wichita, Kansas
  - Central Kentucky Research Associates Inc., Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Centex Studies Inc., Lake Charles, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Regional Urology LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - BTC of New Bedford, New Bedford, Massachusetts
  - Regeneris Medical, North Attleboro, Massachusetts
  - Infinity Medical Research Inc., North Dartmouth, Massachusetts
  - Beacon Clinical Research, Quincy, Massachusetts
  - Bay State Clinical Trials Inc., Watertown, Massachusetts
  - Remidica LLC, Rochester, Michigan
  - Saginaw Valley Medical Research, Saginaw, Michigan
  - CentraCare Clinic Adult & Pediatric Urology, Sartell, Minnesota
  - Poplar Bluff Urology, Poplar Bluff, Missouri
  - Montana Health Research Institute Inc., Billings, Montana
  - Montana Medical Research, Missoula, Montana
  - Pioneer Clinical Research, LLC, Bellevue, Nebraska
  - Barrett Clinic P.C., La Vista, Nebraska
  - Women's Clinic of Lincoln PC, Lincoln, Nebraska
  - Meridian Clinical Research LLC, Norfolk, Nebraska
  - Adult and Pediatric Urology P.C., Omaha, Nebraska
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research Consortium, Las Vegas, Nevada
  - Sheldon Freedman MD Ltd, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Premier Urology Group LLC, Edison, New Jersey
  - Urologic Research and Consulting LLC, Englewood, New Jersey
  - Lawrence OB-GYN Clinical Research LLC, Lawrenceville, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - AccumetRx Clinical Research - Division of Urology Group of New Mexico, Albuquerque, New Mexico
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research Inc., Endwell, New York
  - AccuMed Research Associates, Garden City, New York
  - Drug Trials America, Hartsdale, New York
  - Smart Medical Research Inc., Jackson Heights, New York
  - ProHealth Care AssociatesLLP, Port Jefferson, New York
  - Rochester Clinical Research Inc., Rochester, New York
  - Upstate Clinical Research Associates LLC, Williamsville, New York
  - PMG Research of Cary, Cary, North Carolina
  - PMG Research of Charlotte LLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Raleigh Medical Group PMG Research of Raleigh, Raleigh, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research, Wilmington, North Carolina
  - Carolina Medical Trials LLC, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Sentral Clinical Research Services, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Buckeye Health and Research, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Providence Health Partners, Dayton, Ohio
  - HWC Womens Research Center, Englewood, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Family Practice Center of Wadsworth Inc. - New Venture Medical Research, Wadsworth, Ohio
  - Ohio Clinical Research LLC, Willoughby Hills, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Leonard Maliver MD Antria, Inc., Indiana, Pennsylvania
  - The Clinical Trial Center LLC, Jenkintown, Pennsylvania
  - Green and Seidner Family Practice Associates P.C., Lansdale, Pennsylvania
  - Clinical Research of Philadelphia LLC, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians Inc., Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists Hills ObGyn Associates Inc, Pittsburgh, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians Inc., Uniontown, Pennsylvania
  - PEAK Research LLC, Upper Saint Clair, Pennsylvania
  - Greater Providence Clinical Research, LLC, East Providence, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Pharmacorp Clinical Trials Inc., Charleston, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - DeGarmo Institute of Medical Research, Greer, South Carolina
  - PMG Research of Charleston LLC, Moncks Corner, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Charleston LLC, Mt. Pleasant, South Carolina
  - Family Medicine of SayeBrook LLC, Myrtle Beach, South Carolina
  - Palmetto Institute of Clinical Research Inc., Pelzer, South Carolina
  - Hillcrest Clinical Research LLC, Simpsonville, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - PMG Research of Bristol LLC, Bristol, Tennessee
  - WR - ClinSearch LLC, Chattanooga, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - MultiSpecialty Clinical Research, Inc., Johnson City, Tennessee
  - Volunteer Research Group - NOCCR, Knoxville, Tennessee
  - Adams Patterson Gynecology and Obstetrics, Memphis, Tennessee
  - Clinical Research Associates Inc., Nashville, Tennessee
  - DiscoveResearch Inc., Bryan, Texas
  - WR Global Medical Research, DeSoto, Texas
  - Advances in Health, Houston, Texas
  - Centex Studies Inc., Houston, Texas
  - Discovery MM Services Inc., Houston, Texas
  - BI Research Center, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Discovery MM Services Inc., Katy, Texas
  - Discovery MM Services Inc., Missouri City, Texas
  - Village Health Partners ACRC Trials, Plano, Texas
  - Clinical Trials of Texas Inc., San Antonio, Texas
  - Bandera Family Health Care, San Antonio, Texas
  - Clinova Clinical Trials, Spring, Texas
  - Progressive Clinical Research, Bountiful, Utah
  - Wasatch Clinical Research LLC, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Millennium Clinical Trials, Arlington, Virginia
  - Health Research of Hampton Roads Inc., Newport News, Virginia
  - Seattle Urology Research, Burien, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - North Spokane Womens Health, Spokane, Washington
- Canada (7):
  - Central Alberta Research Clinic, Red Deer, Alberta
  - Silverado Research Inc., Victoria, British Columbia
  - PrimeHealth Clinical Research, Toronto, Ontario
  - Manna Research (Quebec), Lévis, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Manna Research (Montreal), Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Hungary (5):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Szarka Ödön Egyesitett Egeszsegügyi es Szocialis Intezmeny, Csongrád
  - Szent Anna Private Surgery, Debrecen
  - Mediroyal Prevention Center, Kecskemét
  - Uro-clin Ltd, Pécs
- Latvia (3):
  - Daugavpils Regional Hospital, Daugavpils
  - Uro Ltd., Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (3):
  - Public Institution Republican Klaipda Hospital, Klaipėda
  - Vilnius, Vilnius
  - Vilnius city Clinical hospital, Vilnius
- Poland (6):
  - Poradnia Urologiczna EuroMediCare Szpital Specjalistyczny z Przychodnia, Wroclaw, Woj. Dolnoslaskie
  - ETG Lodz, Lodz, Woj. Lodzkie
  - NZOZ NOVITA Specjalistyczne Gabinety Lekarskie, Lublin, Woj. Lubelskie
  - Nzoz Heureka, Piaseczno, Woj. Mazowieckie
  - Klimed Marek Klimkiewicz, Bialystok, Woj. Podlaskie
  - NZOZ Centrum Urologiczne sp. z o.o., Mysłowice, Woj. Slaskie

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staskin D, Frankel J, Gregg SG, Varano S, Owens-Grillo J. Plain language summary of safety and symptom improvement with vibegron in people with overactive bladder: results from the EMPOWUR study. J Comp Eff Res. 2023 Sep;12(9):CER. doi: 10.57264/cer-2023-0043. Epub 2023 Aug 10. PMID 37586057
- [Derived] Frankel J, Staskin D, Varano S, Newman DK, Gregg SG, Owens-Grillo J. Plain language summary: does treatment with vibegron result in improvements in overactive bladder (OAB) symptoms that are meaningful to people with OAB? J Comp Eff Res. 2023 Sep;12(9):CER. doi: 10.57264/cer-2023-0049. Epub 2023 Aug 10. PMID 37586052
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- [Derived] Newman DK, Thomas E, Greene H, Haag-Molkenteller C, Varano S. Efficacy and Safety of Vibegron for the Treatment of Overactive Bladder in Women: A Subgroup Analysis From the Double-Blind, Randomized, Controlled EMPOWUR Trial. Urogynecology (Phila). 2023 Jan 1;29(1):48-57. doi: 10.1097/SPV.0000000000001258. Epub 2022 Oct 21. PMID 36384907
- [Derived] Staskin D, Frankel J, Varano S, Kennelly M, Newman DK, Rosenberg MT, Shortino DD, Jankowich RA, Mudd PN Jr. Vibegron for the Treatment of Patients with Dry and Wet Overactive Bladder: A Subgroup Analysis from the EMPOWUR Trial. Int J Clin Pract. 2022 Apr 13;2022:6475014. doi: 10.1155/2022/6475014. eCollection 2022. PMID 35685566
- [Derived] Frankel J, Staskin D, Varano S, Kennelly M, Newman DK, Rosenberg MT, Jankowich RA, Shortino D, Mudd PN Jr, Girman CJ. Interpretation of the Meaningfulness of Symptom Reduction with Vibegron in Patients with Overactive Bladder: Analyses from EMPOWUR. Adv Ther. 2022 Feb;39(2):959-970. doi: 10.1007/s12325-021-01972-8. Epub 2021 Dec 18. PMID 34921665
- [Derived] Varano S, Staskin D, Frankel J, Shortino D, Jankowich R, Mudd PN Jr. Efficacy and Safety of Once-Daily Vibegron for Treatment of Overactive Bladder in Patients Aged >/=65 and >/=75 Years: Subpopulation Analysis from the EMPOWUR Randomized, International, Phase III Study. Drugs Aging. 2021 Feb;38(2):137-146. doi: 10.1007/s40266-020-00829-z. Epub 2021 Jan 20. PMID 33469832
- [Derived] Frankel J, Varano S, Staskin D, Shortino D, Jankowich R, Mudd PN Jr. Vibegron improves quality-of-life measures in patients with overactive bladder: Patient-reported outcomes from the EMPOWUR study. Int J Clin Pract. 2021 May;75(5):e13937. doi: 10.1111/ijcp.13937. Epub 2021 Jan 22. PMID 33332699

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 3149 participants screened for this study, 1518 were randomized (after a 2-week, single-blind placebo Run-in Period), and 1515 received 1 dose of double-blind study drug in the Treatment Period (Safety Set: placebo, N = 540; vibegron, N = 545; tolterodine, N = 430).
Groups:
- Placebo: Participants received matching placebo, orally, once daily for 12 weeks. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- Vibegron 75 mg: Participants received vibegron 75 milligrams (mg), orally, once daily for 12 weeks. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- Tolterodine ER 4 mg: Participants received tolterodine extended release (ER) 4 mg, orally, once daily for 12 weeks. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
Period: Overall Study
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Started | 540 | 547 | 431
Completed | 486 | 502 | 385
Not Completed | 54 | 45 | 46
Not completed — Withdrawal by Subject | 21 | 14 | 13
Not completed — Lost to Follow-up | 14 | 15 | 10
Not completed — Adverse Event | 6 | 8 | 13
Not completed — Lack of Efficacy | 3 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 3
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawn Due to Sponsor | 1 | 0 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Captured as Other in Database | 8 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data are reported for members of the Safety Set, comprised of all participants who received at least 1 dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg | Total
Number analyzed (Participants) | 540 | 545 | 430 | 1515
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (13.35) | 60.4 (13.49) | 59.8 (13.27) | 60.0 (13.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 459 | 463 | 364 | 1286
  Male | 81 | 82 | 66 | 229
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska | 3 | 2 | 0 | 5
  Asian | 30 | 28 | 27 | 85
  Black or African American | 85 | 78 | 72 | 235
  White | 418 | 435 | 326 | 1179
  Puerto Rican | 1 | 1 | 1 | 3
  White and Black or African American | 1 | 0 | 0 | 1
  Hispanic | 2 | 1 | 0 | 3
  Filipino | 0 | 0 | 1 | 1
  Morrocan | 0 | 0 | 1 | 1
  Multiracial | 0 | 0 | 1 | 1
  White, Black or African American | 0 | 0 | 1 | 1
Average number of micturitions per 24 hours in all overactive bladder (OAB) participants [Mean (Standard Deviation); unit: micturitions per 24 hours] — A micturition/void was defined as "Urinated in Toilet" as indicated on the Patient Voiding Diary (PVD). The number of micturitions was defined as the number of times a participant voided in the toilet as indicated on the PVD. The average daily number of micturitions was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of micturitions that occurred on a Complete Diary Day (CDD) divided by the number of CDDs in the PVD. Population: Only participants with available data were analyzed.
  micturitions per 24 hours
    number analyzed (Participants) | 537 | 544 | 430 | 1511
    (all) | 11.72 (3.971) | 11.38 (3.508) | 11.53 (3.184) | 11.54 (3.595)
Average number of urge urinary incontinence (UUI) episodes per 24 hours in OAB Wet participants [Mean (Standard Deviation); unit: UUI episodes] — The number of UUI episodes was defined as the number of times a participant had checked "urge" as the main reason for the leakage in the PVD, regardless of whether more than one reason for leakage in addition to "urge" was checked. OAB Wet participants were those participants with an average of ≥8.0 micturitions per Diary Day (DD); with an average of ≥1.0 UUI episodes per DD; and, if stress urinary incontinence was present, with a total number of UUI episodes greater than the total number of stress urinary incontinence episodes from the previous visit diary. Population: Only participants with available data were analyzed.
  UUI episodes
    number analyzed (Participants) | 537 | 544 | 430 | 1511
    (all) | 2.80 (2.978) | 2.78 (3.105) | 2.72 (2.616) | 2.77 (2.926)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (CFB) at Week 12 in the Average Number of Micturitions Per 24 Hours in All Overactive Bladder (OAB) Participants
Description: A micturition/void is defined as "Urinated in Toilet" as indicated on the Patient Voiding Diary (PVD). The number of micturitions is defined as the number of times a participant voided in the toilet as indicated on the PVD. The average daily number of micturitions was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of micturitions that occurred on a Complete Diary Day (CDD) divided by the number of CDDs in the PVD. CFB was calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD). Covariates included in the mixed model for repeated measures are study visit (Weeks 2, 4, 8, and 12), OAB type (wet/dry), sex, region (U.S./non-U.S.), BL number of micturitions, and treatment by study visit interaction. FAS=Full Analysis Set.
Time Frame: Baseline (BL); Week 12
Population: FAS: all randomized participants who took at least 1 dose of double-blind study treatment and had at least 1 evaluable CFB measurement. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: micturitions per 24 hours
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 475 | 492 | 378
micturitions per 24 hours | -1.3 (0.14) | -1.8 (0.14) | -1.6 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.001, Mixed Model for Repeated Measures (MMRM) — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.2], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0988, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.16

2. Primary Outcome: CFB at Week 12 in the Average Number of Urge Urinary Incontinence (UUI) Episodes Per 24 Hours in OAB Wet Participants
Description: The number of UUI episodes is defined as the number of times a participant had checked "urge" as the main reason for the leakage in the PVD, regardless of whether more than one reason for leakage in addition to "urge" was checked. The average daily number of UUI episodes was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of UUI episodes that occurred on a CDD divided by the number of CCDs in the PVD. CFB was calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when participant got up for the day each morning and time participant got up for the day the next morning as recorded in the PVD). Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), sex, region (U.S./non-U.S.), BL number of UUI episodes and treatment by study visit interaction. FAS-I=Full Analysis Set for Incontinence.
Time Frame: Baseline; Week 12
Population: FAS-I: all randomized OAB Wet participants who took at least 1 dose of double-blind study treatment and had at least 1 evaluable CFB measurement. Only those participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: UUI episodes per 24 hours
Groups:
- Placebo: OAB Wet: Participants who met the definition of OAB Wet at study entry (based on the PVD) received matching placebo, orally, once daily for 12 weeks. OAB Wet participants were defined as those with an average of ≥8.0 micturitions per Diary Day; with an average of ≥1.0 UUI episodes per Diary Day; and, if stress urinary incontinence was present, with a total number of UUI episodes greater than the total number of stress urinary incontinence episodes from the previous visit diary. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- Vibegron 75 mg: OAB Wet: Participants who met the definition of OAB Wet at study entry (based on the PVD) received vibegron 75 milligrams (mg), orally, once daily for 12 weeks. OAB Wet participants were defined as those with an average of ≥8.0 micturitions per Diary Day; with an average of ≥1.0 UUI episodes per Diary Day; and, if stress urinary incontinence was present, with a total number of UUI episodes greater than the total number of stress urinary incontinence episodes from the previous visit diary. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
- Tolterodine ER 4 mg: OAB Wet: Participants who met the definition of OAB Wet at study entry (based on the PVD) received tolterodine extended release (ER) 4 mg, orally, once daily for 12 weeks. OAB Wet participants were defined as those with an average of ≥8.0 micturitions per Diary Day; with an average of ≥1.0 UUI episodes per Diary Day; and, if stress urinary incontinence was present, with a total number of UUI episodes greater than the total number of stress urinary incontinence episodes from the previous visit diary. Participants were stratified by Baseline Overactive Bladder Type (Wet versus Dry) and sex.
Arm/Group | Placebo: OAB Wet | Vibegron 75 mg: OAB Wet | Tolterodine ER 4 mg: OAB Wet
Number analyzed (Participants) | 372 | 383 | 286
UUI episodes per 24 hours | -1.4 (0.13) | -2.0 (0.13) | -1.8 (0.14)
Statistical Analysis 1: Comparison: Placebo: OAB Wet vs Vibegron 75 mg: OAB Wet; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.3], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo: OAB Wet vs Tolterodine ER 4 mg: OAB Wet; Test type: Superiority; p = 0.0123, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.7 to -0.1], Standard Error of Mean 0.15

3. Secondary Outcome: CFB at Week 12 in the Average Number of Urgency Episodes Over 24 Hours in All OAB Participants
Description: An urgency episode is defined as the "Need to Urinate Immediately" as indicated on the PVD. CFB is calculated as the post-BL value minus the BL value. "Over 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD). Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), OAB type (wet/dry), sex, region (U.S./non-U.S.), BL number of urgency episodes, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: urgency episodes over 24 hours
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 475 | 492 | 378
urgency episodes over 24 hours | -2.0 (0.19) | -2.7 (0.19) | -2.5 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p = 0.0020, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-1.1 to -0.2], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0648, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -0.4, 95% CI 2-sided [-0.9 to 0.0], Standard Error of Mean 0.23

4. Secondary Outcome: Percentage of OAB Wet Participants With at Least a 75% Reduction From Baseline in UUI Episodes Per 24 Hours at Week 12
Description: The number of UUI episodes is defined as the number of times a participant had checked "urge" as the main reason for the leakage in the PVD, regardless of whether more than one reason for leakage in addition to "urge" was checked. The average daily number of UUI episodes was calculated using the daily entries in the PVD (which was to be completed prior to each study visit) as the total number of UUI episodes that occurred on a CDD divided by the number of CCDs in the PVD. CFB was calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when participant got up for the day each morning and time participant got up for the day the next morning as recorded in the PVD).
Time Frame: Baseline; Week 12
Population: FAS-I. The multiple imputation method was used for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: OAB Wet | Vibegron 75 mg: OAB Wet | Tolterodine ER 4 mg: OAB Wet
Number analyzed (Participants) | 405 | 403 | 319
percentage of participants
  Unadjusted | 36.8 | 52.4 | 47.6
  Adjusted for sex | 32.8 | 49.3 | 42.2
Statistical Analysis 1: Comparison: Placebo: OAB Wet vs Vibegron 75 mg: OAB Wet; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel risk difference estimate was stratified by sex (female/male), with weights proposed by Greenland and Robins; Difference in percentage = 16.5, 95% CI 2-sided [9.7 to 23.4]
Statistical Analysis 2: Comparison: Placebo: OAB Wet vs Tolterodine ER 4 mg: OAB Wet; Test type: Superiority; p = 0.0120, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Difference in percentage = 9.4, 95% CI 2-sided [2.1 to 16.7]

5. Secondary Outcome: Percentage of OAB Wet Participants With a 100% Reduction From Baseline in UUI Episodes Per 24 Hours at Week 12
Description: as for outcome 4
Time Frame: Baseline; Week 12
Population: FAS-I. The multiple imputation method was used for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: OAB Wet | Vibegron 75 mg: OAB Wet | Tolterodine ER 4 mg: OAB Wet
Number analyzed (Participants) | 405 | 403 | 319
percentage of participants
  Unadjusted | 22.5 | 28.8 | 26.6
  Adjusted for sex | 19.0 | 25.3 | 20.9
Statistical Analysis 1: Comparison: Placebo: OAB Wet vs Vibegron 75 mg: OAB Wet; Test type: Superiority; p = 0.0360, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Difference in percentage = 6.3, 95% CI 2-sided [0.4 to 12.1]
Statistical Analysis 2: Comparison: Placebo: OAB Wet vs Tolterodine ER 4 mg: OAB Wet; Test type: Superiority; p = 0.5447, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Difference in percentage = 1.9, 95% CI 2-sided [-4.1 to 7.8]

6. Secondary Outcome: Percentage of All OAB Participants With at Least a 50% Reduction From Baseline in Urgency Episodes Per 24 Hours at Week 12
Description: An urgency episode is defined as the "Need to Urinate Immediately" as indicated on the PVD. CFB is calculated as the post-BL value minus the BL value. "Per 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD).
Time Frame: Baseline; Week 12
Population: FAS. The multiple imputation method was used for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 520 | 526 | 417
percentage of participants
  Unadjusted | 38.3 | 43.2 | 41.2
  Adjusted for sex | 32.8 | 39.5 | 36.4
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p = 0.0235, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel risk difference estimate was stratified by sex and OAB type (wet/dry), with weights proposed by Greenland and Robins; Difference in percentage = 6.8, 95% CI 2-sided [0.9 to 12.7]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.2400, Cochran-Mantel-Haenszel; [statistical method as in outcome 6, analysis 1]; Difference in percentage = 3.7, 95% CI 2-sided [-2.5 to 10.0]

7. Secondary Outcome: CFB at Week 12 in the Average Number of Total Incontinence Episodes Over 24 Hours in OAB Wet Participants
Description: Total incontinence is defined as having any reason for "Accidental Urine Leakage" and/or "Accidental Urine Leakage" checked, as indicated on the PVD. It is assumed that if the participant recorded a reason for leakage then the accidental urine leakage occurred. CFB is calculated as the post-BL value minus the BL value. "Over 24 hours" corresponds to one Diary Day (i.e., time between when the par. got up for the day each morning and time the par. got up for the day the next morning as recorded in the PVD). Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), sex, region (U.S./non-U.S.), BL number of incontinence episodes, and treatment by study visit interaction. hr = hours.
Time Frame: Baseline; Week 12
Population: FAS-I. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: total incontinence episodes over 24 hr
Arm/Group | Placebo: OAB Wet | Vibegron 75 mg: OAB Wet | Tolterodine ER 4 mg: OAB Wet
Number analyzed (Participants) | 372 | 383 | 286
total incontinence episodes over 24 hr | -1.6 (0.15) | -2.3 (0.15) | -2.0 (0.16)
Statistical Analysis 1: Comparison: Placebo: OAB Wet vs Vibegron 75 mg: OAB Wet; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-1.0 to -0.4], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Placebo: OAB Wet vs Tolterodine ER 4 mg: OAB Wet; Test type: Superiority; p = 0.0074, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.8 to -0.1], Standard Error of Mean 0.17

8. Secondary Outcome: CFB at Week 12 in the Coping Score From the Overactive Bladder Questionnaire Long Form (OAB-q LF, 1-week Recall) in All OAB Participants
Description: The OAB-q LF is a validated patient-reported outcome. 8 questions of the OAB-q LF ask participants how well they have coped with their bladder symptoms during the previous week, as a measure of quality of life. Each question has a response ranging from "not coping" (= 1) to "coping well" (= 6). These questions make up the coping scale. The raw score (sum of question scores [ranging from 8 to 48]) is transformed to a unified score, ranging from 0 to 100. Higher scores correspond to a higher quality of life, and lower scores represent a lower quality of life. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), sex, region (U.S./non-U.S.), OAB type (wet/dry), BL score, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with evaluable data were analyzed. If < 50% of items were available, the subscore was regarded as missing; however, if ≥ 50% of items were available, the subscore included missing items imputed as the average of the remaining non-missing items for the subscore.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 504 | 512 | 400
units on a scale | 12.9 (1.32) | 16.5 (1.31) | 16.0 (1.39)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p = 0.0039, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = 3.6, 95% CI 2-sided [1.2 to 6.0], Standard Error of Mean 1.24
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0210, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = 3.1, 95% CI 2-sided [0.5 to 5.7], Standard Error of Mean 1.32

9. Secondary Outcome: CFB at Week 12 in the Average Volume Voided Per Micturition in All OAB Participants
Description: A micturition/void is defined as "Urinated in Toilet" as indicated on the PVD. The number of micturitions is defined as the number of times a participant voided in the toilet as indicated on the PVD. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), OAB type (wet/dry), sex, region (U.S./non-U.S.), BL volume (milliliters [mL]), and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL per micturition
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 478 | 490 | 375
mL per micturition | 2.2 (3.28) | 23.5 (3.26) | 15.5 (3.52)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = 21.2, 95% CI 2-sided [14.3 to 28.1], Standard Error of Mean 3.52
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p < 0.001, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = 13.3, 95% CI 2-sided [5.9 to 20.7], Standard Error of Mean 3.76

10. Secondary Outcome: CFB at Week 12 in the Health-related Quality of Life (HRQL) Total Score From the OAB-q LF (1-week Recall) in All OAB Participants
Description: The OAB-q LF is a validated patient-reported outcome. The 25 questions comprising the Coping, Concern, Sleep and Social Interaction subscales of the OAB-q LF ask participants how much their symptoms have affected their life over the last week. Each question has a response ranging from "None of the time" (= 1) to "All of the time" (= 6). The raw score (sum of question scores for the 4 subscales [ranging from 25 to 150]) is transformed to a unified score, ranging from 0 to 100. Higher scores correspond to a higher quality of life, and lower scores represent a lower quality of life. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), sex, region (U.S./non-U.S.), OAB type (wet/dry), BL score, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 504 | 512 | 400
units on a scale | 10.8 (1.13) | 14.6 (1.12) | 13.7 (1.19)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = 3.8, 95% CI 2-sided [1.7 to 5.8], Standard Error of Mean 1.06
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0114, MMRM; Least Squares Mean Difference = 2.9, 95% CI 2-sided [0.6 to 5.1], Standard Error of Mean 1.13

11. Secondary Outcome: CFB at Week 12 in the Symptom Bother Score From the OAB-q LF (1-week Recall) in All OAB Participants
Description: The OAB-q LF is a validated patient-reported outcome. The first 8 questions of the OAB-q LF ask participants how much they were bothered by their bladder symptoms during the previous week. Each question has a response ranging from "Not at all" (= 1) to "A very great deal" (= 6). These questions make up the symptom bother scale. The raw score (sum of question scores [ranging from 8 to 48]) is transformed to a unified score, ranging from 0 to 100. Higher scores correspond to the symptoms having a larger bother, and lower scores represent a lower amount of bother due to symptoms. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), sex, region (U.S./non-U.S.), OAB type (wet/dry), BL score, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 504 | 512 | 400
units on a scale | -12.8 (1.25) | -19.6 (1.24) | -17.4 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -6.9, 95% CI 2-sided [-9.2 to -4.6], Standard Error of Mean 1.17
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p < 0.001, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -4.6, 95% CI 2-sided [-7.1 to -2.2], Standard Error of Mean 1.25

12. Secondary Outcome: Percentage of All OAB Participants With an Average Number of Micturitions < 8 Per 24 Hours at Week 12
Description: A micturition/void is defined as "Urinated in Toilet" as indicated on the PVD. The number of micturitions is defined as the number of times a participant voided in the toilet as indicated on the PVD. A participant was defined as having an average of < 8 daily micturitions if the arithmetic mean of the number of micturitions per day in the PVD was less than 8 . "Per 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD).
Time Frame: Week 12
Population: FAS. Only participants with evaluable data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 520 | 526 | 417
percentage of participants
  Unadjusted | 28.7 | 40.1 | 35.0
  Adjusted for sex | 24.8 | 37.2 | 31.6
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — CMH=Cochran-Mantel-Haenszel; The CMH risk difference estimate was stratified by OAB type (wet/dry) and sex (female/male), with weights proposed by Greenland and Robins; Difference in percentage = 12.4, 95% CI 2-sided [6.7 to 18.1]
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0236, Cochran-Mantel-Haenszel; [statistical method as in outcome 12, analysis 1]; Difference in percentage = 6.9, 95% CI 2-sided [0.9 to 12.8]

13. Secondary Outcome: Percentage of OAB Wet Participants With at Least a 50% Reduction From Baseline in Total Incontinence Episodes Per 24 Hours at Week 12
Description: Total incontinence is defined as having any reason for "Accidental Urine Leakage" and/or "Accidental Urine Leakage" checked, as indicated on the PVD. It is assumed that if the participant recorded a reason for leakage then the accidental urine leakage occurred. All events marked as having leakage, regardless of cause, or where "Accidental Leakage" was checked. were used in the analysis. "Per 24 hours" corresponds to one Diary Day (i.e., time between when the participant got up for the day each morning and time the participant got up for the day the next morning as recorded in the PVD.
Time Frame: Baseline; Week 12
Population: FAS-I. Only participants with evaluable data were analyzed. The multiple imputation method was used for missing values.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo: OAB Wet | Vibegron 75 mg: OAB Wet | Tolterodine ER 4 mg: OAB Wet
Number analyzed (Participants) | 405 | 403 | 319
percentage of participants
  Unadjusted | 53.8 | 64.0 | 66.5
  Adjusted for sex | 49.9 | 61.6 | 61.5
Statistical Analysis 1: Comparison: Placebo: OAB Wet vs Vibegron 75 mg: OAB Wet; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Difference in percentage = 11.7, 95% CI 2-sided [4.7 to 18.6]
Statistical Analysis 2: Comparison: Placebo: OAB Wet vs Tolterodine ER 4 mg: OAB Wet; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel; [statistical method as in outcome 4, analysis 1]; Difference in percentage = 11.5, 95% CI 2-sided [4.2 to 18.9]

14. Secondary Outcome: CFB at Week 12 in Overall Bladder Symptoms Based on Patient Global Impression of Severity (PGI-Severity) in All OAB Participants
Description: The Patient Global Impression (PGI) questions are designed to assess a participant's overall impression of OAB. For the PGI-Severity score, participants are asked to rate their OAB symptoms over the previous week with one of the following responses: 1 = none, 2 = mild, 3 = moderate, 4 = severe. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), OAB type (wet/dry), sex, region (U.S./non-U.S.), BL score, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 484 | 494 | 382
units on a scale | -0.5 (0.04) | -0.8 (0.04) | -0.7 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.04
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p = 0.0055, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.1, 95% CI 2-sided [-0.2 to 0.0], Standard Error of Mean 0.05

15. Secondary Outcome: CFB at Week 12 in Overall Control Over Bladder Symptoms Based on Patient Global Impression of Control (PGI-Control) in All OAB Participants
Description: The Patient Global Impression (PGI) questions are designed to assess a participant's overall impression of OAB. For the PGI-Control score, participants were asked to rate how much control they had over their OAB symptoms over the previous week with one of the following responses: 1 = complete control, 2 = a lot of control, 3 = some control, 4 = only a little control, 5 = no control. CFB is calculated as the post-BL value minus the BL value. Covariates included in the mixed model for repeated measures were study visit (Weeks 2, 4, 8, and 12), OAB type (wet/dry), sex, region (U.S./non-U.S.), BL score, and treatment by study visit interaction.
Time Frame: Baseline; Week 12
Population: FAS. Only participants with evaluable data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
Number analyzed (Participants) | 484 | 494 | 382
units on a scale | -0.7 (0.05) | -1.0 (0.05) | -0.9 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Vibegron 75 mg; Test type: Superiority; p < 0.0001, MMRM — Hypothesis testing was performed for vibegron minus placebo; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.4 to -0.2], Standard Error of Mean 0.05
Statistical Analysis 2: Comparison: Placebo vs Tolterodine ER 4 mg; Test type: Superiority; p < 0.001, MMRM — Comparisons between tolterodine ER and placebo are considered descriptive; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.3 to -0.1], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: from the time the participant provided informed consent to participate in the study at the Screening Visit until completion of the Follow-up Visit (up to Day 113 or Early Withdrawal plus 28 days)
Description: Treatment-emergent adverse events are reported for members of the Safety Set, comprised of all participants who received at least 1 dose of study treatment. Participants were included in the treatment group corresponding to the study treatment they actually received for the analysis of safety data.
Arm/Group | Placebo | Vibegron 75 mg | Tolterodine ER 4 mg
All-Cause Mortality (participants affected / at risk) | 0/540 | 0/545 | 1/430
Serious Adverse Events (participants affected / at risk) | 6/540 | 8/545 | 10/430
Other Adverse Events (participants affected / at risk) | 38/540 | 36/545 | 50/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=540) | Vibegron 75 mg (N=545) | Tolterodine ER 4 mg (N=430)
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=540) | Vibegron 75 mg (N=545) | Tolterodine ER 4 mg (N=430)
Dry mouth (Gastrointestinal disorders) | 5 | 9 | 28
Urinary tract infection (Infections and infestations) | 33 | 27 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor does not object to publication by Institution or Principal Investigator (PI) of results of the Trial based on information collected or generated by the Institution or PI. However, the Institution and PI are required to provide the Sponsor with an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed to ensure against any inadvertent disclosure of Sponsor Confidential Information or unprotected Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03492281/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT03492281/SAP_001.pdf